CLINICAL TRIAL: NCT02604862
Title: Exploratory Clinical Study to Image the Intrapulmonary Microdosing of FIBroproliferation ONE (FIB ONE) Using Endomicroscopy
Brief Title: Imaging FIB ONE in the Human Lung Using Endomicroscopy
Acronym: FIB ONE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FIB ONE
Record Dates: First submitted 2015-11-09; First posted 2015-11-16 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Fibrosis; Lung Cancer
MeSH Terms: conditions — Fibrosis; Lung Neoplasms | interventions — 4-((5-chloro-2-pyridinyl)oxy)-1-((((4S)-4-methyl-2,5-dioxo-4-imidazolidinyl)methyl)sulfonyl)-piperidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FIB ONE administration (Experimental): All participants in this clinical study will be dosed on one occasion with FIB ONE. The final dosage will be less than 100 µg.
  Interventions: Other: FIB ONE; Other: AZD1236
- AZD1236 administration (Experimental): To quantify the change in mean FIB ONE fluorescence amplification gradient in the presence of AZD1236 in the fibroproliferative lung
  Interventions: Other: FIB ONE; Other: AZD1236

INTERVENTIONS:
Other: FIB ONE — FIB ONE will be administered to each patient during a bronchoscopy procedure. Fibre-based endomicroscopy and two types of viewer software will be used to detect FIB ONE signal in the lung.
Other: AZD1236 — AZD1236 will be delivered at microdose concentrations and is thus considered to be unable to exert any pharmacologic effect outside the area of administration and unlikely to cause an adverse reaction.

SUMMARY:
While the process of fibrosis is essential for normal wound healing, an excessive and uncontrolled 'fibrotic' response can result in impaired tissue structure and function. In other words, affected 'fibrotic' tissues are unable to heal back to normal and therefore don't work as effectively as they normally would.

In the case of the lung, fibrosis can occur across large parts of the lung such as in conditions like Idiopathic Pulmonary Fibrosis (IPF) and sarcoidosis or it can occur in much smaller patches such as around the borders of some lung tumours. At the moment the investigators don't fully understand the mechanisms of fibrosis and so therefore cannot monitor or treat these conditions as effectively as the investigators could. Despite the significant global financial burden of these diseases, treatment options are very limited and monitoring of disease progression remains a real challenge.

In an effort to address this problem, the research group are currently developing a library of novel optical molecular imaging SmartProbes that are targeted against key pathological processes in the human lung. The functional profile for this portfolio of probes is that they exhibit high stability and specificity in vivo and have a short activation time permitting rapid point-of-care in situ molecular profiling enabling in the future, improved diagnostic certainty and stratification for targeted pharmacological intervention. This clinical microdosing study protocol focuses around the intrapulmonary delivery of microdoses (<100µg) of the Smartprobe Fibroproliferation (FIB ONE) to disparate regions of the human lung to highlight MMP activity combined with an active MMP inhibitor (AZD1236) to the distal lung. This approach will enable the research team to directly demonstrate the utility of this SmartProbe-based platform in the validation of drug target engagement in areas of suspected fibroproliferation (characterised by increased MMP activity).

DETAILED DESCRIPTION:
The primary endpoint is to visualise the delivery of a microdose of FIB ONE and assess imaging parameters in patients with lung conditions using two microendoscopy systems (Part A). A secondary objective is to quantify the change in mean FIB ONE fluorescence amplification gradient in the presence of AZD1236 in the fibroproliferative lung (Part B). Imaging will be performed using a novel multi-colour widefield fluorescence microendoscopy platform and a commercially available imaging platform.

Cohort 1 will consist of 20 patients scheduled for routine elective diagnostic or surveillance bronchoscopy with a fibroproliferative lung condition and Cohort 2 will consist of 6 patients undergoing planned cardiothoracic surgery for biopsy/resection of lung conditions characterised by excessive activity of the fibroproliferative pathway. For both cohorts, eligibility will be verified by a clinical trial physician after written informed consent has been obtained.

For cohort 1, a bronchoscopy with lavage will be performed to harvest broncho-alveolar lavage fluid (BALF). For cohort 2, a sample of resected lung tissue will be analysed. Fibre-based endomicroscopy (FE) will be performed and up to 100μg of FIB ONE and PBS/AZD1236 will be instilled. CT identified regions of architecturally normal lung in all participants will act as internal controls and will be used to compare MMP activity in normal and diseased lung tissue.

Participants will be asked to provide routine blood samples before and after FIB ONE and AZD1236 administration. A cardiorespiratory exam and routine observations will be performed 4-6 hours following administration and all participants will be assessed for discharge. All participants will either be contacted by a member of the research team via telephone or ward visit 24 hours (± 4 hours) after dosing to ensure no AEs/SAEs were experienced. The participant's involvement in the study is concluded when the 24 hour assessment has been successfully completed and all AEs/SAEs have been resolved.

ELIGIBILITY:
Inclusion Criteria:

All Cohorts Capacity to provide informed consent

* ≥ 16 years
* Attending consultant permission for bronchoscopy
* Thoracic CT scan taken within the previous 10 weeks
* Readily accessible target areas with bronchoscopy and FE
* Cohort 1 - Patients with a suspected or confirmed lung condition associated with increased activity of the fibroproliferative pathway and scheduled to undergo an elective bronchoscopy
* Cohort 2 - Patients undergoing planned cardiothoracic surgery for biopsy/resection of a lung condition associated with increased activity of the fibroproliferative pathway.

Exclusion Criteria:

* All Cohorts
* Refusal for participation by attending consultant
* Any history of anaphylaxis
* Significant coagulopathy or bleeding tendency, which causes bronchoscopy to be unsuitable, as determined by clinical co-investigator or the participant's attending consultant, using information which is routinely available
* Myocardial infarction in the preceding four weeks
* Women who are pregnant or are breastfeeding
* Receiving drugs that cause increased autofluorescence in the lung, specifically amiodorane and methotrexate

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
The measurement of FIB ONE fluorescence intensity in the lung (Part A). | Analysis to take one week to complete post procedure.
  Quantify the change in fluorescence upon delivery of FIB ONE.

SECONDARY OUTCOMES:
The measurement of FIB ONE fluorescence intensity in the lung in the presence of PBS or AZD1236 (Part B). | Analysis to take one week to complete post procedure.
  Quantify the change in fluorescence upon delivery of FIB ONE and AZD1236/PBS.

CONTACTS AND LOCATIONS:
Overall Officials: Kev Dhaliwal, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No